CLINICAL TRIAL: NCT06637371
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Integrated Single Ascending Dose, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 691 in Healthy Participants and Participants With Mild-to-Moderate Asthma
Brief Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study Evaluating AMG 691 in Healthy Participants and Participants With Mild-to-Moderate Asthma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20230151
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: AMG 691; Pulmonology; Immunology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (Experimental): Healthy participants will be randomized in a 3:1 ratio to receive either AMG 691 or placebo.
  Interventions: Drug: AMG 691; Drug: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Healthy participants will be randomized in a 3:1 ratio to receive either AMG 691 or placebo.
  Interventions: Drug: AMG 691; Drug: Placebo
- Part C: Multiple Dose (Experimental): Participants with mild-to-moderate asthma will be randomized in a 2:1 ratio to receive either AMG 691 or placebo.
  Interventions: Drug: AMG 691; Drug: Placebo

INTERVENTIONS:
Drug: AMG 691 — Subcutaneous (SC) injection
Drug: Placebo — SC injection

SUMMARY:
The main objective of this study is to assess the safety and tolerability of AMG 691 as single doses (healthy participants only) and multiple doses in healthy participants and participants with mild-to-moderate asthma.

ELIGIBILITY:
Inclusion Part A and B

* Participants must be capable of giving informed consent and have provided informed consent.
* Participants must be 18 to 65 inclusive at time of signing of informed consent.
* Participants must have a Body Mass Index between 18.0 to 30 kg/m2 and total body weight ≥ 40 kg at screening.
* Participants must be overtly healthy as determined by the investigator based on medical evaluation and study screening procedures.
* Female participants must be of non-childbearing potential.

Inclusion Part C

* Participants must be capable of giving informed consent and have provided informed consent.
* Participants must be 18 to 65 inclusive at time of signing of informed consent.
* Participants must have documentation of physician diagnosed asthma for ≥ 12 months prior to screening.
* Participants must have documented bronchodilator responsiveness of forced expiratory volume in 1 second (FEV1) ≥ 12% and ≥200 mL in the 10 years before screening or at the screening visit.
* Participants must have a pre-bronchodilator percent predicted FEV1 between 50 and 100% inclusive at screening visit and Day -1.
* Participants must have peripheral blood eosinophils ≥ 200 cells/μl at screening visit and Day -1
* Participants must have a fractional exhaled nitric oxide (FeNO) ≥ 25 ppb at screening visit and Day -1.
* Participant must not use inhaled corticosteroids (ICS) or must be treated with low-dose or medium-dose ICS and on a stable dose for a minimum of 12 weeks prior to screening.

Exclusion (applicable to all study parts)

* History of malignancy (except for in situ cervical cancer or surgically excised non-melanoma skin cancer occurring more than 5 years prior to randomization).
* History of anaphylaxis or hypersensitivity to biologic therapy or sensitivity to mammalian derived products.
* History of immunodeficiency or history of severe infection within the last 3 years requiring IV antibiotics.
* History of tuberculosis (TB), TB symptoms, or positive interferon gamma release assay.
* History of untreated or unresolved helminthic infection within 24 weeks of day 1.
* Positive human immunodeficiency virus (HIV) antibodies, hepatitis B core antigen, hepatitis B core antibody, or hepatitis C virus (HCV) ribonucleic acid (RNA).
* Male participants unwilling to follow contraceptive requirements.

Additional Exclusion for Part C only

* Female of childbearing potential not willing to use 2 methods of contraception with one being a highly effective method of contraception.
* History of pulmonary disease that may interfere with interpretation of study results.
* History of upper respiratory infection within 6 weeks of screening.
* Asthma Control Questionnaire (ACQ-6) > 3
* Asthma symptoms or exacerbations requiring 2 or more systemic corticosteroid bursts (≥10 mg/day prednisone or equivalent for ≥ 3 days each) in the previous 12 months.
* More than one hospitalization or emergency department visit in the last year.
* History of life-threatening asthma exacerbation requiring admission to intensive care unit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately 11 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. Serious AEs (SAEs) are defined as any untoward medical occurrence that, meet at least 1 of the following serious criteria: Immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect. Includes AEs of interest (AEOI), and AEs leading to discontinuation.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of AMG 691 | Up to approximately 11 months
Area Under the Curve (AUC) of AMG 691 | Up to approximately 11 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- United States (10):
  - Orange County Research Center, Lake Forest, California
  - Translational Clinical Research LLC, Aventura, Florida
  - Destiny Research Center, Palmetto Bay, Florida
  - ClinCept, LLC, Columbus, Georgia
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - University of North Carolina Clinical and Translational Research Center, Chapel Hill, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Endeavor Clinical Trials, San Antonio, Texas
- Clinical Medical and Analytical eXellence CMAX, Adelaide, South Australia, Australia
- Algemeen Ziekenhuis Sint Maarten-Emmaus vzw, Mechelen, Belgium
- Winchester District Memorial Hospital, Winchester, Ontario, Canada
- United Kingdom (3):
  - VPD Heart and Lung Research Institute, Cambridge
  - Chelsea and Westminster Hospital, London
  - The Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com